CLINICAL TRIAL: NCT05436522
Title: Effects of Total Intravenous Anesthesia With Remimazolam vs Propofol on Intraoperative Hypotension in Major Noncardiac Surgery: a Randomized Controlled Trial
Brief Title: REmimazolam vs PrOpofol on Intraoperative hypotenSion in Major Noncardiac surgEry
Acronym: REPOSE-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFEC-2021-260
Record Dates: First submitted 2022-05-09; First posted 2022-06-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Intraoperative Hypotension
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam TIVA (Experimental): Induction: Remimazolam, sufentanil, cisatracurium. Maintenance: Remimazolam, remifentanil, cisatracurium.
  Interventions: Drug: Remimazolam
- Propofol TIVA (Active Comparator): Induction: Propofol, sufentanil, cisatracurium. Maintenance: Propofol, remifentanil, cisatracurium.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is administered intravenously for induction and maintenance of general anesthesia. The dose is titrated to maintain Bispectral Index value between 40 and 60.
  Arms: Remimazolam TIVA
Drug: Propofol — Propofol is administered intravenously for induction and maintenance of general anesthesia. The dose is titrated to maintain Bispectral Index value between 40 and 60.
  Arms: Propofol TIVA

SUMMARY:
Intraoperative hypotension is common during major noncardiac surgery and is associated with adverse postoperative outcomes. Propofol, the most commonly used intravenous anesthetic agent worldwide, is associated with hypotension on induction and maintenance of general anesthesia. Remimazolam is a newly developed short-acting benzodiazepine drug and has been approved for use in procedural sedation and general anesthesia. It was associated with a lower incidence of hypotension during procedural sedation in previous studies. The aim of this study is to tested the primary hypothesis that total intravenous anesthesia with remimazolam reduces the duration and severity of hypotension during major noncardiac surgery compared with total intravenous anesthesia with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years;
* Undergoing elective major surgery under general anesthesia (expected surgery time >2 h, expected length of postoperative stay >2 d);
* Need for intraoperative invasive blood pressure monitoring via arterial line;
* Fulfilling ≥1 of the following criteria (a-k):

  1. history of coronary artery disease;
  2. history of stroke;
  3. history of congestive heart failure;
  4. preoperative NT-proBNP >200 pg/mL;
  5. preoperative high sensitivity troponin T > 14 ng/L;
  6. age ≥70 years;
  7. diabetes requiring medical treatment;
  8. ASA status 3 or 4;
  9. history of chronic kidney disease (preoperative sCr >133μmol/L or 1.5 mg/dL);
  10. preoperative serum albumin <30 g/L;
  11. preoperative hemoglobin <100 g/L.

Exclusion Criteria:

* Undergoing organ transplantation, cardiac, neurological, or adrenal gland surgery;
* Planned intraoperative MAP higher or lower than 65 mmHg;
* Severe untreated or uncontrolled hypertension (preoperative SBP >180 mmHg and/or DBP >110 mmHg);
* End-stage renal disease requiring renal-replacement therapy;
* ASA score ≥5;
* Preoperative requirement of vasopressor infusion;
* Unable to receive bispectral index monitoring;
* Known allergy to benzodiazepines, propofol, opioids or cisatracurium;
* Current participation in another interventional study;
* Previous participation in this study;
* Pregnant or breastfeeding women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Time-weighted average (TWA) intraoperative mean arterial pressure (MAP) under 65 mmHg. | MAP measurements are recorded every minute from of anesthesia induction to end of wound closure.
  TWA-MAP under 65 mmHg for each patient is derived by dividing area under the curve (AUC)-MAP under 65 mmHg by the time interval between the first and the last MAP measurements.

SECONDARY OUTCOMES:
AUC-MAP under 65 mmHg. | From of anesthesia induction to end of wound closure.
  AUC-MAP under 65 mmHg for each patient is derived by depth of hypotension in millimeters of mercury below a MAP of 65 mmHg × time in minutes spent below a MAP of 65 mmHg.
Duration of MAP under 65 mmHg. | From of anesthesia induction to end of wound closure.
  Duration of MAP under 65 mmHg is the total amount of time in minutes that the MAP is under 65 mmHg.
Time-weighted average (TWA) intraoperative mean arterial pressure (MAP) under 70 mmHg. | From of anesthesia induction to end of wound closure.
  TWA-MAP under 70 mmHg for each patient is derived by dividing area under the curve (AUC)-MAP under 70 mmHg by the time interval between the first and the last MAP measurements.
AUC-MAP under 70 mmHg. | From of anesthesia induction to end of wound closure.
  AUC-MAP under 70 mmHg for each patient is derived by depth of hypotension in millimeters of mercury below a MAP of 70 mmHg × time in minutes spent below a MAP of 70 mmHg.
Duration of MAP under 70 mmHg. | From of anesthesia induction to end of wound closure.
  Duration of MAP under 70 mmHg is the total amount of time in minutes that the MAP is under 70 mmHg.
Time-weighted average (TWA) intraoperative mean arterial pressure (MAP) under 60 mmHg. | From of anesthesia induction to end of wound closure.
  TWA-MAP under 60 mmHg for each patient is derived by dividing area under the curve (AUC)-MAP under 60 mmHg by the time interval between the first and the last MAP measurements.
AUC-MAP under 60 mmHg. | From of anesthesia induction to end of wound closure.
  AUC-MAP under 60 mmHg for each patient is derived by depth of hypotension in millimeters of mercury below a MAP of 60 mmHg × time in minutes spent below a MAP of 60 mmHg.
Duration of MAP under 60 mmHg. | From of anesthesia induction to end of wound closure.
  Duration of MAP under 60 mmHg is the total amount of time in minutes that the MAP is under 60 mmHg.
Postoperative complications. | From end of surgery to 30 days after surgery.
  A composite of in-hospital all-cause mortality and cardiovascular, neurological, renal, respiratory, and infectious complications.
Days alive and at home. | From end of surgery to 30 days after surgery.
  Number of days alive and at home within 30 days after surgery.
Postoperative quality of recovery. | At postoperative day 1.
  Patient-reported quality of recovery after surgery and anesthesia with the QoR-15, ranging from 0 (poor recovery) to 150 (excellent recovery)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
The deidentified IPD will be shared upon reasonable request after study completion.